CLINICAL TRIAL: NCT01055990
Title: Phase1 An Observational Clinical Trial With an Influenza A (H1N1) 2009 Monovalent,Split-virion Vaccine in Healthy Adults, Aged 18-60 Years Phase2 Basic and Clinical Research on Applying Blood Fix to Treat Critical H1N1 Patients
Brief Title: Basic and Clinical Research on Applying Blood Fix to Treat Critical H1N1 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Collaborators: Beijing Ditan Hospital (Other); National Institute for the Control of Pharmaceutical and Biological Products, China (Other)
Responsible Party: Lu Hong-zhou, Shanghai Public Health Clinical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-0015
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2009-11

CONDITIONS: Virus Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza; Orthomyxoviridae Infections
Keywords: pandemic influenza A (H1N1) 2009; blood fix treatment; influenza A (H1N1) 2009 monovalent vaccine; effectiveness; immunogenicity; safety
MeSH Terms: conditions — Virus Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heathy,aged 18-60 years, (Other): They are healthy, are 18-60 years of age, did not have a history of infection with the 2009 H1N1 virus, and are appropriate to vaccination, without any interdictions. And they guardians confirmed that they understood the study procedures, provided written informed consent, and agreed to comply with the following visit schedule. Woman participants all are not pregnant,with a negative pregnancy test before vaccination.
  Interventions: Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg
- clinically critical H1N1 patients (Experimental): The critical H1N1 patients as recipients whose conditions are confirmed according to current standard for critical H1N1 diagnosis. The study wll research H1N1 viral load in blood of critical H1N1 patients and swab nucleic acid testing parallelity; measure H1N1 viral Load in blood and swabs (adopting Real-time PCR method) of 5 to 10 victims; and the planned blood taking time is the tenth day since the fever begins.
  Interventions: Other: blood fix

INTERVENTIONS:
Biological: split-virion, non-adjuvanted H1N1 vaccine of 15 μg — The influenza A (H1N1) 2009 monovalent, (Split-virion)inactivated vaccine was developed by Shanghai Institute of Biological Products, and the seed virus was prepared from reassortant vaccine virus A/California/7/2009,distributed by the Centers for Disease Control and Prevention in the United States. This strain was recommended by the World Health Organization and obtained from the Chinese Food and Drug Administration.The vaccine adopted the assessment of experts, and formally accessed to the approval document number of production and new drug certificate issued by the Chinese Food and Drug Administration.
  Arms: Heathy,aged 18-60 years,
Other: blood fix — The blood fix with a hemagglutination-inhibition titer of 1:80 or more than was collected from healthy persons who are inoculated with specific H1N1 vaccine
  Arms: clinically critical H1N1 patients

SUMMARY:
The 2009 flu pandemic is a global outbreak of a new strain of influenza A virus subtype H1N1, commonly known as swine flu, that was first identified in April 2009. Large-scale immunization is an essential approach of controlling the pandemic.Vaccines are now becoming available for protection against pandemic influenza A(H1N1) 2009 infection in some countries.In response to the pandemic, novel vaccines against the virus strain A/California/07/2009(H1N1) have been developed and recently were approved for vaccination among specific populations in China. However, the safety and effectiveness of the vaccines is of prime concern to the authorities and the public.This report details the findings of a observational clinical trial of the safety and immunogenicity of a influenza A (H1N1)2009 monovalent vaccine.

The virus of Swine Flu H1N1 that outbroke in 2009 is sensitive to neuraminidase inhibitors (Oseltamivir, zanamivir and peramivir) but have drug resistant to adamantanamine derivatives (amantadine and Flumadine), therefore neuraminidase inhibitors are recommended for antiviral therapy against Swine Flu H1N1, effect of which is evidence by the data that such drugs do modify the symptoms and decrease the death rate of H1N1 in America and Mexico. However, clinically, the investigators have encountered that this virus can infect resistant strains of Oseltamivir, which urges for a more effective treatment plan.

In view of above situations, seeking for an effective measures against H1N1 flu should be a top priority and will benefit human life and economy globally. This Topic will take the classic strategy of passive immunity to perform basic and clinical researches on applying blood fix to treat critical H1N1 patients and collect blood of healthy persons who are inoculated with specific H1N1 vaccines to cure critical H1N1 patients.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization (WHO) to declare a pandemic on June 11, 2009. Antiviral drugs, such as oseltamivir or zanamivir, may be effective in treating cases of swine flu, but large-scale immunization is an essential approach of controlling the pandemic.Although preliminary evidence from a matched case-control study suggests some protection from the 2008-9 trivalent inactivated vaccine against pandemic influenza A/H1N1 2009, particularly severe forms of the disease. A vaccine against H1N1 is expected to be the most effective tool for controlling influenza A (H1N1) infection.In response to the pandemic, novel vaccines against the virus strain A/California/07/2009(H1N1) have been developed and recently were approved for vaccination among specific populations in China.The primary safety objective of this study is to assess the safety of split- virion inactivated H1N1 vaccine without adjuvant when administered at the 15 ug dose.The primary immunogenicity objective is to assess the hemagglutinin antibody and neutralizing antibody response following split- virion inactivated A(H1N1) vaccine without adjuvant. Participants 148 healthy persons age 18-60 years who have no history of novel influenza H1N1 2009 infection or novel influenza H1N1 2009 vaccination. This is an observational, Phase II study in healthy males and non-pregnant females, aged 18-60 years.This study is designed to investigate the safety and immunogenicity of an inactivated influenza H1N1 virus vaccine after approved by the Chinese Food and Drug Administration.Following immunization, safety will be measured by assessment of adverse events through 21 days. Immunogenicity testing will be hemagglutination inhibition (HI) assays and microneutralization (MN) assays on serum obtained on the day 0,7 and 21 after vaccination.In addition, we will take clinical researches on applying blood fix to treat critical H1N1 patients and collect blood of healthy persons who are inoculated with H1N1 vaccines to cure critical H1N1 patients and further observe the effectiveness and safety, for the purpose of working out a new weapon against H1N1. According to the Blood Donation Law of the People's Republic of China, the blood donation shall follow principle of voluntary.The donors should be healthy persons inoculated with specific H1N1 vaccine and their titer of H1N1 hemagglutination inhibition antibody must be 1：320 or more than after examination (the kit shall be provided by the WHO) by Shanghai Municipal Center for Disease Control and Prevention.

ELIGIBILITY:
Inclusion Criteria:

phase 1：

1. Healthy male or female aged 18-60 years
2. Volunteers are able to understand and sign the informed consent
3. Be able to show legal identity card for the sake of recruitment
4. Voluntarily receive a dose of influenza A (H1N1) 2009 monovalent vaccine - phase 2: 1)The donors :Healthy male or female aged 18-60 years; inoculated with specific H1N1 vaccine; titer of H1N1 hemagglutination inhibition antibody must be 1:80 or more than after examination (the kit shall be provided by the WHO) by Shanghai Municipal Center for Disease Control and Prevention 2)The patients: clinical H1N1patients with positive swab nucleic acid Real-time PCR test; critical H1N1 patients;fever less than 10 days;virus viremia was Preferred

Exclusion Criteria:

phase 1:

1. Cases or cured cases of influenza A (H1N1) virus infection
2. Women of pregnancy, lactation or about to be pregnant in recency
3. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
4. Autoimmune disease or immunodeficiency
5. Guillain-Barre Syndrome
6. Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen
7. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
8. Axillary temperature > 37.0 centigrade at the time of dosing
9. Uncontrolled epilepsy, and other progressive neurological diseases
10. Suffering from acute illness, serious chronic diseases, acute exacerbation of chronic diseases and flu
11. Administration of any other investigational research agents within 30 days before the dosing
12. Any other reasons that health care giver consider inappropriate to vaccination, and so on phase 2: 1)The donors :Do not meet donation requirements;the titer of H1N1 hemagglutination inhibition antibody less than 1:80 2)The patients:clinically mild H1N1 patients; fever more than 10 days;Clinicians believe that the patient was not suitable for blood fix treatment and so on

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-04 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
apply blood fix to treat critical H1N1 patients and further observe the effectiveness and safety, for the purpose of working out a new weapon against H1N1 | 30 minutes ahead of blood transfusion,6 hours, 12 hours, 24 hours and 48 hours after transfusion

SECONDARY OUTCOMES:
Hemagglutination inhibition antibody titer and Microneutralization antibody titer | D0,D7,D21
local and systemic adverse reaction after vaccination | Day1-21

CONTACTS AND LOCATIONS:
Overall Officials: Hong-zhou Lu, Professor, Study Director — Fudan University
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Zhu FC, Wang H, Fang HH, Yang JG, Lin XJ, Liang XF, Zhang XF, Pan HX, Meng FY, Hu YM, Liu WD, Li CG, Li W, Zhang X, Hu JM, Peng WB, Yang BP, Xi P, Wang HQ, Zheng JS. A novel influenza A (H1N1) vaccine in various age groups. N Engl J Med. 2009 Dec 17;361(25):2414-23. doi: 10.1056/NEJMoa0908535. Epub 2009 Oct 21. PMID 19846844
- [Background] Wu J, Fang HH, Chen JT, Zhou JC, Feng ZJ, Li CG, Qiu YZ, Liu Y, Lu M, Liu LY, Dong SS, Gao Q, Zhang XM, Wang N, Yin WD, Dong XP. Immunogenicity, safety, and cross-reactivity of an inactivated, adjuvanted, prototype pandemic influenza (H5N1) vaccine: a phase II, double-blind, randomized trial. Clin Infect Dis. 2009 Apr 15;48(8):1087-95. doi: 10.1086/597401. PMID 19281330
- [Background] Greenberg ME, Lai MH, Hartel GF, Wichems CH, Gittleson C, Bennet J, Dawson G, Hu W, Leggio C, Washington D, Basser RL. Response to a monovalent 2009 influenza A (H1N1) vaccine. N Engl J Med. 2009 Dec 17;361(25):2405-13. doi: 10.1056/NEJMoa0907413. Epub 2009 Sep 10. PMID 19745216
- [Background] Clark TW, Pareek M, Hoschler K, Dillon H, Nicholson KG, Groth N, Stephenson I. Trial of 2009 influenza A (H1N1) monovalent MF59-adjuvanted vaccine. N Engl J Med. 2009 Dec 17;361(25):2424-35. doi: 10.1056/NEJMoa0907650. Epub 2009 Sep 10. PMID 19745215
- [Derived] Sun F, Zhang Y, Tian D, Zheng M, Liu L, Zhang R, Dai Z, Chen J, Li T, Lu H. Responses after one dose of a monovalent influenza A (H1N1) 2009 inactivated vaccine in Chinese population--a practical observation. Vaccine. 2011 Sep 2;29(38):6527-31. doi: 10.1016/j.vaccine.2011.07.006. Epub 2011 Jul 19. PMID 21767595
- See also: Click here for more information about this disease:The Pandemic influenza A (H1N1) 2009 — http://www.nlm.nih.gov/medlineplus/flu.html
- See also: Related Info — http://clinicaltrials.gov/ct2/info/fdalinks